CLINICAL TRIAL: NCT07142291
Title: A Phase IIB Randomized, Double-Blind, Placebo-Controlled, Multi-Dose Study to Evaluate the Effects of PHENOGENE-1A (Cromolyn) as an Adjuvant Treatment in Subjects With Mild to Moderate Amyotrophic Lateral Sclerosis (ALS)
Brief Title: PHENOGENE-1A (Cromolyn) Treatment in Patients With Mild to Moderate ALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PhenoNet, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHENOALS-001
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; Lou Gehrigs Disease; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Cromolyn Sodium; BID protein, human; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose PHENOGENE-1A (17.1 mg BID) (Experimental): 17.1 mg, BID, oral inhalation via dry powder inhaler
  Interventions: Drug: Cromolyn Sodium (17.1 mg BID); Drug: Riluzole (100 mg)
- High Dose PHENOGENE-1A (34.2 mg BID) (Experimental): 34.2 mg, BID, oral inhalation via dry powder inhaler
  Interventions: Drug: Cromolyn Sodium (34.2 mg BID); Drug: Riluzole (100 mg)
- Placebo (Placebo Comparator): Placebo comparator matched to active treatment, BID, oral inhalation via dry powder inhaler
  Interventions: Drug: Placebo; Drug: Riluzole (100 mg)

INTERVENTIONS:
Drug: Cromolyn Sodium (34.2 mg BID) — 17.1 mg, BID, oral inhalation
  Other Names: Cromolyn; Sodium Cromoglycate
  Arms: High Dose PHENOGENE-1A (34.2 mg BID)
Drug: Cromolyn Sodium (17.1 mg BID) — 34.2 mg, BID, oral inhalation via dry powder inhaler
  Other Names: Cromolyn; Sodium Cromoglycate; PHENOGENE-1A
  Arms: Low Dose PHENOGENE-1A (17.1 mg BID)
Drug: Placebo — Placebo comparator matched to active treatment.
  Arms: Placebo
Drug: Riluzole (100 mg) — 50 mg, oral tablet, BID, standard of care treatment
  Other Names: Rilutek

SUMMARY:
The purpose of this study is to test the effects of PHENOGENE-1A, which is the treatment under investigation in this study. This research will investigate if PHENOGENE-1A can help people with ALS by measuring their function using the ALS Functional Rating Scale Revised (ALSFRS-R), measuring lung function using pulmonary function tests (PFTs), such as forced vital capacity (FVC), and measuring neuro-inflammatory biomarkers in the blood.

DETAILED DESCRIPTION:
This is a Phase IIB, randomized, double-blind, placebo-controlled study designed to assess the effects of PHENOGENE-1A (oral inhalation via dry powder inhaler [DPI]) in subjects with mild to moderate ALS disease. Eligible subjects will be randomized to receive either low dose PHENOGENE-1A (34.2 mg per day: in 2 doses of 17.1 mg and matching placebo BID), high dose PHENOGENE-1A (68.4 mg per day: 34.2 mg BID), or placebo (2 matching placebo capsules BID) (see table below), in a 2:2:1 ratio. Subjects will receive treatment for a duration of 24 weeks. All subjects must be on a stable dose of Riluzole 50 mg BID (100 mg daily) for at least 4 weeks prior to randomization and must continue their Riluzole regimen, 50 mg BID (100 mg daily), as standard-of-care treatment, throughout the 24 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ALS; the diagnosis of ALS defined by revised El Escorial criteria as follows:

   1. Evidence of lower motor neuron (LMN) degeneration by clinical, electrophysiological, or neuropathological examination.
   2. Evidence of upper motor neuron (UMN) degeneration by clinical examination.
   3. Progressive spread of symptoms or signs within a region or to other regions, as determined by clinical examination or the history of disease progression.
   4. Absence of electrophysiological, neuroimaging, or pathological evidence of other diseases that might explain the UMN or LMN degeneration and exclusion of other causes.
2. Male or female subjects aged 18 to 75 years inclusive.
3. Must provide written informed consent for study-related procedures.
4. Must be capable of completing all study-related procedures, assessments, and visits in the judgment of Investigator.
5. Disease duration from ALS symptom onset of motor weakness ≤24 months.
6. ALSFRS-R total score ≥38 at screening visit.
7. ALSFRS-R Breathing subscore should be ≥9 at the time of screening.
8. ALSFRS-R Bulbar subscore should be ≥9 at the time of screening.
9. Forced vital capacity >70% of predicted value.
10. PIFR ≥100 L/minute.
11. Must be receiving a stable dose of standard-of-care treatment Riluzole for 4-weeks before signing informed consent.
12. Female subjects who are of childbearing potential must agree to use of highly effective methods of contraception consistent with local regulations during the study, and for 3 months after the study drug administration. Examples include the following, but not limited to:

    1. Combined (estrogen and progestogen containing) or progestogen-only hormonal contraceptives;
    2. Intrauterine device or intrauterine hormone-releasing system; OR
    3. Post-menopausal status must have experienced their last menstrual period minimum of 1 year prior to study drug administration; OR
    4. Surgically sterilized. Female subject should be willing to not donate egg during the trial and for 3 months after the last dose of the study drug.
13. Male subjects who are sexually active with a female of childbearing potential must agree to use highly effective contraception as described above, or a combination of 2 acceptable methods of contraception (e.g., a barrier method along with a female partner using a hormonal contraceptive method), in accordance with local regulations, throughout the duration of the study, and for 3 months after the last dose of the study drug.

(Male subject should be willing to not donate sperm during the trial and for 3 months after the last dose of the study drug.)

Exclusion Criteria:

1. ALSFRS-R score change (decrease) by 2.5 or more points between the screening visit and Day 1 (baseline) score.
2. Bulbar onset ALS (<9 bulbar subscore)
3. Any use of non-invasive ventilation (e.g., continuous positive airway pressure, non-invasive bi-level positive airway pressure or non-invasive volume ventilation) for any portion of the day, or mechanical ventilation via tracheostomy, or on any form of oxygen supplementation.
4. Any other significant neurological disorder which can interfere with study assessments, e.g., significant cognitive impairment and/or clinical dementia.
5. Significant psychiatric illness like schizophrenia, bipolar disorder etc. Subjects with depression can be included, only if the depression has been stable and no episode of major depression has occurred in the past year.
6. Severe cardiac disease (e.g., QTc>500 ms), Torsade de Pointes, evidence of significant heart failure (New York Heart Association [NYHA] Class 3 or greater, myocardial infarction or unstable angina in the 6 months prior to screening).
7. Any moderate-to-severe pulmonary disease or difficulty taking inhaled drugs.
8. Inability to tolerate the administration of an oral inhaled powder via DPI.
9. Has taken any investigational product within 30 days or 5 half lives of the drug, whichever is longer, prior to dosing.
10. Taking inhaled protein products on a chronic basis (such as insulin, parathyroid hormone, etc).
11. Subjects with a body weight of 32 kg or less, or a body mass index of <17.5 or >35.0 at time of screening.
12. Moderate-to-severe liver disease: aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3 times the upper limit of normal; total bilirubin > 1.5 x ULN.; subjects with hepatic diseases such as hepatic cirrhosis, hepatic cancer and active hepatitis.
13. Moderate-to-severe renal disease: creatinine clearance <45 mL/min/1.73 m2 (by Cockcroft-Gault calculation).
14. Any clinically significant disorder or laboratory abnormality that, in the Investigator's opinion, could interfere with the subject's participation in the study, place the subject at increased risk, or confound interpretation of the study results.
15. Pregnant or breast-feeding females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Absolute change in ALSFRS-R total score from baseline to Week 24 | Baseline to Week 24
  To evaluate the effects of PHENOGENE-1A (cromolyn) on functional changes in subjects with mild to moderate ALS using the ALS Functional Rating Scale-Revised (ALSFRS-R).
Incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline to Week 24
  To evaluate the safety of PHENOGENE-1A following 24 weeks of twice daily (BID) treatment.

SECONDARY OUTCOMES:
Mean rank for CAFS at Week 24 | Baseline to Week 24
  To evaluate the effects of PHENOGENE-1A on function and survival using the Combined Assessment of Function and Survival (CAFS).
Time to event requiring full-time or nearly full-time respiratory support | Randomization to Week 24
  Time from randomization to the first of 7 consecutive days on which permanent assisted ventilation (invasive or non-invasive) was used for >22 hours/day due to ALS progression.
Mean change in percent predicted forced vital capacity (%FVC) from baseline to Week 24 | Baseline to Week 24
  To evaluate the effect of PHENOGENE-1A on respiratory changes.
Mean change in peak inspiratory flow rate (PIFR) from baseline to Week 24 | Baseline to Week 24
  To evaluate changes in PIFR (L/min) during treatment.
Absolute Values and Changes From Baseline in Vital Signs From Baseline to Week 24 by Treatment Arm | Baseline to Week 24
  Vital signs will include:
  * Systolic blood pressure (mmHg)
  * Diastolic blood pressure (mmHg)
  * Pulse rate (beats per minute)
  * Respiratory rate (breaths per minute)
  * Body temperature (°C or °F, as recorded)
  Results will be summarized as:
  * Absolute values for each parameter at each scheduled visit.
  * Changes from baseline at each visit.
  * Summaries will be presented separately by treatment arm.
Number and Percentage of Subjects With Abnormal Clinical Laboratory Values and Changes From Baseline to Week 24 by Treatment Arm | Baseline to Week 24
  Safety laboratory assessments will include hematology, clinical chemistry, coagulation, and urinalysis panels. Each laboratory result will be classified as normal, abnormal (not clinically significant), or abnormal (clinically significant).
  Results will be summarized as: Number and percentage of subjects with abnormal laboratory values at each post-baseline visit, by treatment arm.
  Summary statistics for absolute values and changes from baseline at each visit.
Number and Percentage of Subjects With Abnormal Physical Examination Findings From Baseline to Week 24 by Treatment Arm | Baseline to Week 24
  The physical examination will assess head/neck, eyes, ears, nose/throat, cardiovascular, respiratory, abdominal, musculoskeletal, extremities, and skin systems. Each system will be classified as normal, abnormal (not clinically significant), or abnormal (clinically significant).
  Results will be summarized as the number and percentage of subjects with abnormal findings at each post-baseline visit.
Number and Percentage of Subjects With Abnormal Neurological Examination Findings From Baseline to Week 24 by Treatment Arm | Baseline to Week 24
  The neurological examination will assess mental status, motor function, sensory function, reflexes, and coordination/cerebellar function. Each domain will be classified as normal, abnormal (not clinically significant), or abnormal (clinically significant).
  Results will be summarized as the number and percentage of subjects with abnormal findings at each post-baseline visit.
Number and Percentage of Subjects With Abnormal Electrocardiogram (ECG) Findings From Baseline to Week 24 by Treatment Arm | Baseline to Week 24
  Standard 12-lead ECGs will be performed at protocol-specified visits. Parameters assessed will include:
  * Heart rate: 60-100 beats per minute (bpm)
  * PR interval: 120-200 milliseconds (ms)
  * QRS duration: 70-110 ms
  * QT interval: < 440 ms in men, < 460 ms in women
  * Corrected QT interval (QTcF, Fridericia's formula): < 450 ms in men, < 470 ms in women
  Each ECG result will be classified by the investigator as normal, abnormal (not clinically significant), or abnormal (clinically significant), using these ranges as reference.
  Results will be summarized as the number and percentage of subjects with abnormal ECG findings at each post-baseline visit.
Number and Percentage of Subjects With Suicidal Ideation, Suicidal Behavior, or Self-Injurious Behavior Without Suicidal Intent on the Columbia Suicide Severity Rating Scale (C-SSRS) From Baseline to Week 24 by Treatment Arm | Baseline to Week 24
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be administered at protocol-specified visits to assess suicidal ideation, suicidal behavior, and self-injurious behavior without suicidal intent.
  * Suicidal ideation will be captured using categories 1-5 of the C-SSRS (ranging from passive wish to be dead to active suicidal ideation with plan and intent).
  * Suicidal behavior will be captured using categories 6-10 of the C-SSRS (preparatory acts, aborted attempts, interrupted attempts, and actual attempts).
  * Self-injurious behavior without suicidal intent will be reported separately.
  Results will be summarized as: Number and percentage of subjects with suicidal ideation, suicidal behavior, and self-injurious behavior without suicidal intent, compared between active treatment and placebo arms.
Number and Percentage of Subjects Who Discontinue Study Participation Due to Adverse Events From Baseline to Week 24 | Baseline to Week 24
  The incidence of study discontinuation attributed to treatment-emergent adverse events (TEAEs) will be assessed. Results will be summarized as the number and percentage of subjects who withdraw from the study due to an adverse event, presented separately by treatment arm.

OTHER OUTCOMES:
Change in plasma neuroinflammatory biomarkers from baseline to Week 24 | Baseline (pre-dose) to Week 24
  To evaluate the impact of two different doses of PHENOGENE-1A on neuroinflammation.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - Honor Health Neurology - Bob Bove Neuroscience Institute, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - Sutter Health - California Pacific Medical Center Research Institute, San Francisco, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Lange Neurology, New York, New York
- Thomayer University Hospital - Fakultní Thomayerova nemocnice, Prague, Czechia
- Charité Centrum für Neurologie, Neurochirurgie und Psychiatrie, Berlin, Germany
- Poland (4):
  - Michalski i Partnerzy Lekarze Spółka Partnerska, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Medyczne NeuroProtect (NeuroProtect Medical Center), Warsaw
  - City Clinic Research, Warsaw
- University Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided